CLINICAL TRIAL: NCT00256711
Title: A Randomised, Open Label, Parallel Group, Multi-Centre, Phase II Study of Progression Free Survival Comparing ZD1839 (IRESSA™) (250 MG Tablet) Versus Vinorelbine (30 MG/M2 Infusion) in Chemonaive, Elderly Patients With Locally Advanced (Stage IIIB) or Metastatic (Stage IV) NSCLC
Brief Title: Phase II Iressa Versus Vinorelbine (INVITE)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D791AC00001; INVITE
Record Dates: First submitted 2005-11-20; First posted 2005-11-22 (Estimated); Last update posted 2009-04-23 (Estimated); Status verified 2009-04

CONDITIONS: Non-Small-Cell Lung Carcinoma
Keywords: Locally advanced or metastatic NSCLC.; Stage IIIb or Stage IV lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Gefitinib; Vinorelbine

INTERVENTIONS:
Drug: Gefitinib
Drug: Vinorelbine

SUMMARY:
This is a randomized, open label, parallel group, multi-centre, phase II study of progression free survival, comparing oral ZD1839 (IRESSA™) (250 mg tablet once daily) to vinorelbine 30 mg/m2 infusion on days 1 and 8 of a 21-day cycle) in chemonaïve, elderly patients with locally advanced (stage IIIB) or metastatic (stage IV) non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed NSCLC and willing to provide paraffin embedded tumour tissue
* NSCLC - locally advanced (Stage IIIB) or metastatic (stage IV) disease, not amenable to curative surgery or radiotherapy chemonaïve, life expectancy of 12 weeks
* WHO Performance status <= 2

Exclusion Criteria:

* Newly diagnosed CNS metastases
* Less than 4 weeks since completion of radiotherapy or persistence of any radiotherapy related toxicity.
* Hypersensitivity to ZD1839 or intravenous vinorelbine
* Prior treatment with EGFR inhibitors
* Other co-existing malignancies
* ALT/AST >2.5 x ULRR
* ANC < 2.0 x 10^9/L or platelets < 100 x 10^9/L

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 192
Dates: Start 2004-07; Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
To compare ZD1839 and vinorelbine in terms of progression free survival

SECONDARY OUTCOMES:
To compare ZD1839 and vinorelbine in terms of pulmonary symptom improvement weekly for 18 weeks.
To compare ZD1839 and vinorelbine in terms of quality of life 3 weekly for 18 weeks then 6 weekly.
To compare ZD1839 and vinorelbine in terms of adverse event profile continuous monitoring.
To compare ZD1839 and vinorelbine in terms of overall objective tumour response rate (complete response and partial response) 6 weekly to progression.
To compare ZD1839 and vinorelbine in terms of overall survival (time to death) continuous monitoring

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Iressa Medical Science Director, MD, Study Director — AstraZeneca
Locations (55):
- Australia (5):
  - Research Site, St Leonards, New South Wales
  - Research Site, Westmead, New South Wales
  - Research Site, South Brisbane, Queensland
  - Research Site, Nedlands, Western Australia
  - Research Site, Victoria
- Brazil (4):
  - Research Site, Fortaleza, Ceará
  - Research Site, Goiânia, Goiás
  - Research Site, Rio de Janeiro, Rio de Janeiro
  - Research Site, São Paulo, São Paulo
- Czechia (8):
  - Research Site, Prague, CZ
  - Research Site, Ústí nad Labem, CZ
  - Research Site, Hradec Králové
  - Research Site, Kutná Hora
  - Research Site, Olomouc
  - Research Site, Ostrava
  - Research Site, Ostrava - Poruba
  - Research Site, Pilsen
- France (4):
  - Research Site, Marseille
  - Research Site, Montpellier
  - Research Site, Pierre-Bénite
  - Research Site, Vesoul
- Germany (10):
  - Research Site, Heidelberg, Baden-Wurttemberg
  - Research Site, Ulm, Baden-Wurttemberg
  - Research Site, München, Bavaria
  - Research Site, Hamburg, Hamburg
  - Research Site, Magdeburg, Saxony-Anhalt
  - Research Site, Bad Segeberg, Schleswig-Holstein
  - Research Site, Berlin, State of Berlin
  - Research Site, Großhansdorf
  - Research Site, Halle
  - Research Site, Mainz
- Italy (12):
  - Research Site, La Torretta, Ancona
  - Research Site, Bergamo, BG
  - Research Site, Bologna, BO
  - Research Site, Catania, CT
  - Research Site, Melegnano, MI
  - Research Site, Milan, MI
  - Research Site, Rozzano, MI
  - Research Site, Modena, MO
  - Research Site, Parma, PR
  - Research Site, Orbassano, TO
  - Research Site, Torino, TO
  - Research Site, Napoli
- South Africa (2):
  - Research Site, Cape Town
  - Research Site, Durban
- Research Site, Seoul, South Korea
- Taiwan (2):
  - Research Site, Taichung
  - Research Site, Taipei
- United Kingdom (7):
  - Research Site, Cambridge, Cambrideshire
  - Research Site, Birmingham, West Midlands
  - Research Site, Aberdeen
  - Research Site, Dundee
  - Research Site, Glasgow
  - Research Site, Nottingham
  - Research Site, Sheffield

REFERENCES:
- [Derived] Crino L, Cappuzzo F, Zatloukal P, Reck M, Pesek M, Thompson JC, Ford HE, Hirsch FR, Varella-Garcia M, Ghiorghiu S, Duffield EL, Armour AA, Speake G, Cullen M. Gefitinib versus vinorelbine in chemotherapy-naive elderly patients with advanced non-small-cell lung cancer (INVITE): a randomized, phase II study. J Clin Oncol. 2008 Sep 10;26(26):4253-60. doi: 10.1200/JCO.2007.15.0672. PMID 18779612